CLINICAL TRIAL: NCT02535208
Title: A Pilot Randomized Trial of Restrictive Red Blood Cell Transfusion Guidelines Used in Combination With Near-infrared Spectroscopy Splanchnic-cerebral Oxygenation Ratio Evaluations Versus Liberal Red Blood Cell Transfusion Guidelines in Preterm Infants
Brief Title: Combining Restrictive Guidelines and a NIRS SCORE to Decrease RBC Transfusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-01514
Record Dates: First submitted 2015-08-18; First posted 2015-08-28 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Anemia of Prematurity (AOP)
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive transfusion group (Experimental)
  Interventions: Other: Restrictive transfusions based on SCOR assessment
- Liberal transfusion group (Active Comparator)
  Interventions: Other: Liberal transfusions

INTERVENTIONS:
Other: Restrictive transfusions based on SCOR assessment — RBC transfusions will be given to subjects either when participants' Hgb levels fall below defined values based on respiratory status or, despite not having reached their Hgb trigger threshold, if they manifest symptoms judged by the clinical care team to be consistent with anemia (i.e. apnea, bradycardia, or desaturation episodes) and subsequently have a NIRS evaluation that demonstrates an SCOR < 0.73.
  Arms: Restrictive transfusion group
Other: Liberal transfusions — In the liberal group, RBC transfusions will be given to participants when their Hgb level falls below defined values that are based on respiratory support status, as is standard practice.
  Arms: Liberal transfusion group

SUMMARY:
The primary aim of this study is to determine the mean number of red blood cell (RBC) transfusions received by preterm infants cared for using restrictive Hgb guidelines in combination with splanchnic to cerebral oxygenation ratio (SCOR) assessment compared to the mean number of transfusions received by preterm infants cared for using liberal guidelines alone.

This study is designed as a prospective randomized controlled trial. Preterm infants less than 30 weeks gestational age and 500-1250 grams in weight will be recruited and enrolled into the study during day of life 0 to 3. Study participants will be randomly assigned into two groups: a restrictive transfusion group and a liberal transfusion group. In the liberal group, RBC transfusions will be given to subjects when their Hgb level falls below defined values that are based on respiratory support status. In the restrictive group, RBC transfusions will be given to subjects either when their Hgb level falls below defined values based on respiratory status or, despite not having reached their Hgb trigger threshold, if they manifest symptoms judged by the clinical care team to be consistent with anemia (i.e. apnea, bradycardia, or desaturation episodes) and subsequently have a near-infrared spectroscopy (NIRS) evaluation that demonstrates an SCOR < 0.73.

DETAILED DESCRIPTION:
Previous studies have demonstrated that premature infants transfused using restrictive guidelines, in which red blood cell (RBC) transfusions are triggered at relatively low Hgb thresholds, receive significantly fewer transfusions and have similar clinical outcomes to premature infants transfused using liberal transfusion guidelines that use higher Hgb thresholds. However, some remain apprehensive about a restrictive transfusion approach, primarily because the research remains somewhat limited. In addition, concern also exists because some previous researchers found that although there was no difference in mortality based on whether a restrictive or liberal transfusion guideline was used, they did find that a liberal transfusion policy may provide a neuro-protective benefit. This then implies that there may be circumstances in which a neonate transfused with a restrictive strategy could benefit from an increased Hgb level, but does not receive transfusion because their Hgb has not dropped below a predefined transfusion trigger level.

The investigators have previously demonstrated in an observational study that measuring tissue oxygen saturation (rSO2) levels using near-infrared spectroscopy (NIRS) can be more specific in determining RBC transfusion needs in the preterm population than relying on Hgb values derived from a blood sample. Using a model to calculate the splanchnic to cerebral oxygenation ratio (SCOR) [splanchnic rSO2 / cerebral rSO2] could predict with a high probability if preterm infants would improve clinically after a RBC transfusion. Infants with a low SCOR, who were in a physiologic state in which blood and oxygen were being diverted away from the gastrointestinal tract, usually benefited after transfusion. Neonates with a high SCOR, in which oxygen saturation in gut tissue was relatively constant with brain tissue, were unlikely to improve with transfusion.

The intent of this study is to determine whether the SCOR assessment (performed in addition to traditional measurement of Hbg) can better predict which premature infants will benefit from RBC transfusion in a subset of infants demonstrating signs of anemia before having reached the transfusion threshold of a restrictive transfusion protocol. The goal is to assess whether this additional assessment of oxygen delivery (SCOR) can safely reduce the rate of transfusion in a group of subjects treated on a restrictive protocol compared with those transfused using a liberal transfusion protocol. The hypothesis is that by incorporating a measure of transfusion need, SCOR, to the clinical management of a group of preterm infants following a restrictive guideline approach, we can still reduce the average number of transfusions that these infants receive compared to a similar group of preterm infants managed with a liberal approach, yet have no difference in morbidity, including neurological outcomes.

This study is designed as a prospective randomized controlled trial. Preterm infants less than 30 weeks gestational age and 500-1250 grams in weight will be recruited and enrolled into the study during day of life 0 to 3. Study participants will be randomly assigned into two groups: a restrictive transfusion group and a liberal transfusion group. In the liberal group, RBC transfusions will be given to subjects when their Hgb level falls below defined values that are based on respiratory support status. In the restrictive group, RBC transfusions will be given to subjects either when their Hgb level falls below defined values based on respiratory status or, despite not having reached their Hgb trigger threshold, if they manifest symptoms judged by the clinical care team to be consistent with anemia (i.e. apnea, bradycardia, or desaturation episodes) and subsequently have a near-infrared spectroscopy (NIRS) evaluation that demonstrates an SCOR < 0.73.

ELIGIBILITY:
Inclusion Criteria:

* Inborn patients (NYULMC and Bellevue Hospital) less than or equal to 30 weeks gestational age
* Less than 1250 grams
* Less than 72 hours old at time of parental consent and study inclusion

Exclusion Criteria:

* Preterm neonates with 5 minute Apgar score < 3, 10 minute Apgar score < 5, congenital heart disease, alloimmune hemolytic disease, known chromosomal abnormalities, or major malformations will be excluded.
* Preterm neonates with a birth weight of less than 500 grams will also be excluded
* Any patient already diagnosed with intraventricular hemorrhage (IVH), hydrocephalus or a surgical condition prior to recruitment into the study will be excluded.
* Patients receiving high-frequency ventilation at the time of recruitment will be excluded.
* Any preterm infant who has already received > 2 RBC transfusions prior to enrollment will be excluded.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Average number of RBC transfusions received during neonatal intensive care unit (NICU) stay | Throughout the duration of NICU stay (around 3 months, varies based on infant's overall health)

SECONDARY OUTCOMES:
Presence of common morbidities of prematurity | Throughout the duration of NICU stay (around 3 months, varies based on infant's overall health)
  Common morbidities to be assessed are: Intraventricular hemorrhage (IVH), Periventricular leukomalacia (PVL), Retinopathy of prematurity (ROP), Bronchopulmonary Dysplasia (BPD), and Necrotizing Enterocolitis (NEC)
Difference in growth (weight) between the two groups at various timepoints | At time of NICU dischare (about 3 months), and every 6 months for 3 years
  Investigators will measure differences in both short term and long term physical growth parameters (weight) based upon NICU discharge and return examinations at our NICU follow-up clinic which normally occur every 6 months after discharge for up to 3 years of age.
Difference in growth (length) between the two groups at various timepoints | At time of NICU discharge (about 3 months), and every 6 months for 3 years
  Investigators will measure differences in both short term and long term physical growth parameters (length) based upon NICU discharge and return examinations at our NICU follow-up clinic which normally occur every 6 months after discharge for up to 3 years of age.
Difference in growth (head circumference) between the two groups at various timepoints | At time of NICU discharge (about 3 months), and every 6 months for 3 years
  Investigators will measure differences in both short term and long term physical growth parameters (head circumference) based upon NICU discharge and return examinations at our NICU follow-up clinic which normally occur every 6 months after discharge for up to 3 years of age.
Difference in development between the two groups | When participant reaches 2 years of age
  Developmental outcome will be assessed using the Mullen Scales of Early Learning Test.

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Bailey, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066